CLINICAL TRIAL: NCT02420145
Title: Randomized-controlled Trial of Yoga for Women With Abdominal Obesity
Brief Title: Yoga for Abdominal Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Postdoctoral Researcher, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-6194-BO
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Obesity, Abdominal
MeSH Terms: conditions — Obesity, Abdominal | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): This group will participate in 12 weeks of yoga
  Interventions: Behavioral: Yoga
- Waitlist (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Yoga — 12 weeks of yoga, twice weekly for 90 minutes plus a whole-day workshop
  Arms: Yoga

SUMMARY:
The aim of this randomized trial is to investigate the effects of a 12-week yoga intervention compared to no specific intervention on weight-related outcomes, well-being, and health behaviour in 60 females with abdominal obesity.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference at least 88cm
* Body mass index at least 25
* Sedentary
* Physical and mental ability to participate in the yoga intervention
* Willingness to participate in at least 18 of 24 yoga sessions and the whole-day workshop

Exclusion Criteria:

* Dementia
* Psychosis
* Severe hypertension (diastolic blood pressure more than 120mmHg)
* Type 1 diabetes or insulin-dependent 2 diabetes
* Coronary artery disease
* Myocardial infarction
* Lung embolism
* Stroke
* Regular physical activity or yoga practice
* Pregnancy

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Waist circumference | Week 12

SECONDARY OUTCOMES:
BMI | Week 12
  Body Mass Index
Body weight | Week 12
Quality of life | Week 12
  36-Item Short Form Health Survey (SF-36)
Self esteem | Week 12
  Self-Esteem Scale (SES):
Body awareness | Week 12
  Body Awareness Questionnaire (BAQ)
Body responsiveness | Week 12
  Body Responsiveness Scale (BRS)
Perceived stress | Week 12
  Cohen's Perceived Stress Scale (PSS):
Health-specific self-efficacy | Week 12
  Health-Specific Self-Efficacy Scale
Fruits and vegetables consumption | Week 12
  Five A Day Food Frequency Questionnaire (FADFFQ)
Physical activity | Week 12
  The Questionnaire of Baecke et al. for the Measurement of a Person´s Habitual Physical Activity
Adherence | Week 12
  Class attendance and home practice (log)
Adverse events | Week 12
  Safety will be assessed as adverse events and serious adverse events
Qualitative interview | Week 12
  Qualitative interview on experiences and perceived changes
Waist-hip ratio | Week 12
Bioelectrical impedance analysis | Week 12
Systolic blood pressure | Week 12
Diastolic blood pressure | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen, Essen, Germany